CLINICAL TRIAL: NCT01550536
Title: Aging and Basal Metabolic Rate in Postmenopausal Women: Effects of Long-Term and Short-Term Physical Activity
Brief Title: Physical Activity and Basal Metabolic Rate in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Wenner Gren (Unknown); Sigma Xi (Unknown); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Andrew Froehle, Doctoral Candidate, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UCSD GCRC 1910/6766; 5M01RR000827-35 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Postmenopausal Metabolic Health
Keywords: basal metabolic rate; resting energy expenditure; menopause; physical activity; metabolic syndrome
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Sedentary women who exercised <2 hours per week and who had never engaged in a regular exercise program were enrolled in an exercise training intervention, following baseline measurements. See intervention below.
  Interventions: Behavioral: Resistance and aerobic exercise
- Active (No Intervention): Postmenopausal women who exercised >5 hours per week and had been doing so for at least the past 10 years. These women were asked to maintain their normal activity habits for the duration of the study.

INTERVENTIONS:
Behavioral: Resistance and aerobic exercise — Following baseline measurements, sedentary women were enrolled in a 16-week exercise training program at the YMCA in La Jolla, CA. Exercise occurred 3 times per week, for 1.5 hours each time. Exercise consisted of stretching, 20 minutes of aerobic exercise on elliptical machines, and 3 sets of 10-12 repetitions to failure for each of ten weight lifting exercises: abdominal crunch, arm curl, arm extension, chest press, lat pull-down, leg curl, leg extension, leg press, seated row, and trunk extension. Women started at 65-75% of 1-repetition-maximum, and resistance was increased as necessary to maintain the number of sets and reps and to continue to work to failure. Exercise was monitored by a TechnoGym electronic key system, and trainers instructed and supervised subjects in the gym.
  Arms: Training

SUMMARY:
The primary purpose of this study is to expand research on the effects of physical activity on basal metabolic rate (BMR) in healthy postmenopausal women, and to further compare the effects of long-term habitual exercise to the results of a shorter-term (16 weeks) training program. The investigators will measure BMR by indirect calorimetry and normalize it across subjects for body size (fat free mass) and level of aerobic fitness (VO2MAX). Two groups will be compared: an intervention group (no previous participation in regular exercise, newly enrolled in this study's 16 week training program), and a long-term athlete group (have engaged in at least 5 hours of exercise per week for the past 10 years or longer). A secondary aim is to generate an equation for the prediction of BMR from fat free mass in physically active postmenopausal women, to be applied to hypotheses in biological anthropology. The investigators expect to find at baseline that, controlling for fat free mass and VO2MAX, the long-term group will have significantly higher BMR than the intervention group. At 16 weeks the investigators expect no change in BMR for the long-term group, while BMR will have increased in the intervention group. At the same time, the investigators expect to find that after completing the training regimen, the intervention group will have BMR similar to that of the long-term athletes.

ELIGIBILITY:
Inclusion Criteria:

* naturally postmenopausal (i.e. non-surgically)/> 1 year since last menstruation
* FSH > 30 mIU/ml
* estradiol-17β < 25 pg/ml

Exclusion Criteria:

* smoker, abuser of alcohol/other drugs
* hypo- or hyperthyroid (serum TSH < 0.3 or > 5.5 microU/ml, respectively)
* underweight or severely obese (BMI < 18.5 or > 35 kg/m2, respectively)
* weight instability within the past six months (±> 5% of body weight)
* hormone replacement therapy within the past six months
* history of metabolic, respiratory or cardiovascular disease
* high blood pressure
* contraindication for maximal aerobic testing as determined by PAR-Q questionnaire and physician's examination

Ages: 40 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in basal metabolic rate | baseline, 5, 10 and 16 weeks
  Basal metabolic rate is the energy expended at rest and under fasting conditions.

SECONDARY OUTCOMES:
Change in fat-free mass | baseline, 5, 10 and 16 weeks
Change in maximal aerobic capacity | baseline, 16 weeks
  The maximal oxygen consumption achieved during a graded exercise test to exhaustion. Equipment: electronically-braked cycle ergometer. Participants were screened for CVD risk prior to testing by a physician. Lead II EKG was monitored during testing, and each test was overseen by a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Froehle, PhD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - La Jolla YMCA, La Jolla, California
  - UCSD Human Exercise Physiology Laboratory, La Jolla, California
  - UCSD General Clinical Research Center, San Diego, California

REFERENCES:
- [Result] Froehle AW, Ngo HT, Hopkins SR, Natarajan L, Schoeninger MJ. 2010. Relationship between physical activity, body composition and basal metabolic rate in postmenopausal women. Am J Hum Biol 22:252-253. [meeting abstract]
- [Result] Froehle AW, Ngo HT, Natarajan L, Schoeninger MJ, Hopkins SR. 2011. Short-term exercise does not elevate basal metabolic rate (BMR) in postmenopausal women in the absence of increased fat free mass (FFM). Am J Hum Biol 23:259. [meeting abstract]